CLINICAL TRIAL: NCT00009945
Title: A Clinical Trial Comparing Adjuvant Clodronate Therapy vs Placebo in Early-Stage Breast Cancer Patients Receiving Systemic Chemotherapy and/or Hormonal Therapy or No Therapy
Brief Title: Clodronate With or Without Chemotherapy and/or Hormonal Therapy in Treating Women With Stage I or Stage II Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network); North Central Cancer Treatment Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSABP B-34; SWOG-NSABP-B-34; NCCTG-NSABP-B-34; CDR0000068426
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Clodronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Clodronate (Experimental): Patient receives 2 tablets once daily for 3 years.
  Interventions: Drug: clodronate
- Arm 2: Placebo (Placebo Comparator): Patient receives 2 tablets once daily for 3 years.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: clodronate — 1600 mg PO daily
  Other Names: Bonefos; clodronate disodium
  Arms: Arm 1: Clodronate
Drug: placebo — 2 pills PO daily
  Arms: Arm 2: Placebo

SUMMARY:
RATIONALE: Clodronate may be effective in preventing the spread of cancer to the bones and other parts of the body. It is not yet known whether clodronate is more effective alone or combined with chemotherapy and /or hormonal therapy in preventing metastatic breast cancer.

PURPOSE: Randomized phase III trial to determine the effectiveness of clodronate with or without chemotherapy and /or hormonal therapy in preventing metastases in women who have stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether clodronate administered alone or in addition to adjuvant chemotherapy and/or hormonal therapy improves disease-free survival in women with early stage breast cancer.
* Determine whether clodronate reduces the incidence of skeletal metastases and non-skeletal metastases in these patients.
* Determine whether clodronate improves overall and relapse-free survival in these patients.
* Determine whether clodronate reduces the incidence of skeletal morbidity (e.g., skeletal fractures, hypercalcemia, skeletal pain, need for radiotherapy, spinal cord compression) in these patients.
* Investigate the relevance of serum markers of bone turnover as a prognostic factor for the development of bone metastasis in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified by age (under 50 vs 50 and over), number of positive lymph nodes (0 vs 1-3 vs 4 or more), and hormone receptor status (estrogen receptor [ER] and progesterone receptor [PR] negative vs ER and/or PR positive). Patients are randomized to one of two treatment arms.

Patients in both arms commence treatment within 2 weeks of randomization and continue treatment for 3 years in the absence of bone metastasis or unacceptable toxicity. Study medication must be continued in the case of documented visceral or soft tissue metastasis or other event without skeletal metastasis.

Patients in both arms may also receive adjuvant chemotherapy and/or tamoxifen at the discretion of the protocol investigator. Patients receiving hormonal therapy begin hormonal therapy within 3-12 weeks after the last dose of chemotherapy and continue for a minimum of 5 years.

Patients who have undergone a prior lumpectomy receive adjuvant whole breast radiotherapy. Patients who have undergone a prior mastectomy may receive radiotherapy at the investigator's discretion.

Patients are followed every 6 months for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 3,323 patients will be accrued for this study within 3.5 years.

ELIGIBILITY:
Eligibility

* Patients must have undergone either a total mastectomy or a lumpectomy with either an axillary dissection or sentinel node biopsy. If any sentinel node is histologically positive by H & E, or histologically suspicious on H & E and confirmed positive by immunohistochemistry (IHC), then the patient must have a completion axillary dissection.
* The tumor must be invasive adenocarcinoma on histologic examination with clinical assessment T1-3, N0-1, M0.
* Patients must not be participating in any other clinical trials of systemic therapy for early-stage breast cancer. Patients may participate in the following radiation therapy trials:

  * Node-positive patients may participate in the National Cancer Institute of Canada Clinical Trials Group protocol MA.20, provided the requirements of the B-34 protocol continue to be met. (Node-negative B-34 patients may not participate in MA.20.)
  * Node-positive mastectomy patients may participate in Southwest Oncology Group protocol S9927, provided the requirements of the B-34 protocol continue to be met.
* Patients must have an analysis of both estrogen and progesterone receptors on the primary tumor performed prior to randomization. Tumors will be defined as ER or progesterone receptor (PgR) positive if: 1) the Dextran-coated charcoal or sucrose-density gradient method shows them to have greater than or equal to 10 fmol/mg cytosol protein, or 2) if using individual laboratory criteria they can be shown to be positive by the enzyme immunoassay method (EIA) or immunocytochemical assay. "Marginal or borderline," results (i.e., those not definitively negative) will also be considered positive.
* At the time of randomization, the patient must have had the following within the past 3 months: history and physical exam, a bone scan, thoracic and lumbar spine x-rays, and a chest x-ray. Within the past 12 months patients must have had a gynecologic exam (for women who have a uterus and who will be taking tamoxifen) and a bilateral mammogram.
* At the time of randomization:

  * the postoperative absolute neutrophil count (ANC) must be greater than or equal to 1500/mm3 (or less than 1500/mm3 if, in the opinion of the investigator, this represents an ethnic or racial variation of normal);
  * the postoperative platelet count must be greater than or equal to 100,000;
  * there must be postoperative evidence of adequate hepatic function, i.e.,
  * total bilirubin at or below the upper limit of normal (ULN) for the laboratory; and
  * alkaline phosphatase less than 2.5 x the ULN; and
  * the serum glutamate oxaloacetate transaminase (SGOT)/ aspartate transaminase (AST) less than 1.5 x the ULN;
  * there must be postoperative evidence of adequate renal function (serum creatinine within or less than the laboratory's normal range).
* Serum albumin and serum calcium must be within normal limits.
* A patient with skeletal pain is eligible for inclusion in the study if bone scan and/or roentgenological examination fails to disclose metastatic disease. Suspicious findings must be confirmed as benign by x-ray, MRI, or biopsy.
* Patients with prior nonbreast malignancies are eligible if they have been disease- free for greater than or equal to 5 years before randomization and are deemed at low risk for recurrence by their treating physicians. Patients with squamous or basal cell carcinoma of the skin that has been effectively treated, carcinoma in situ of the cervix that has been treated by surgery only, or lobular carcinoma in situ (LCIS) of the ipsilateral or contralateral breast treated by hormone therapy and/or surgery only are eligible, even if these were diagnosed within 5 years before randomization.
* Patients must have a Zubrod performance status of 0, 1, or 2.
* Special conditions for eligibility of lumpectomy patients: Irradiation and surgery. Patients treated by lumpectomy and axillary node dissection (or no axillary dissection if sentinel node biopsy is negative) to be followed by breast radiation therapy must meet all the eligibility criteria in addition to the following:

  * Generally, lumpectomy should be reserved for tumors less than 5 cm. However, at the investigator's discretion, patients treated with lumpectomy for tumors greater than or equal to 5 cm are eligible.
  * The margins of the resected specimen must be histologically free of invasive tumor and ductal carcinoma in situ (DCIS). For patients in whom pathologic examination demonstrates tumor present at the line of resection, additional operative procedures may be performed to obtain clear margins. This is permissible even if axillary dissection has been performed. Patients in whom tumor is still present at the resected margins after re-excision(s) must undergo total mastectomy to be eligible.

Ineligibility.

* Significant non-malignant bone disease that is likely to interfere with the interpretation of bone x-rays.
* Ulceration, erythema, infiltration of the skin or the underlying chest wall (complete fixation), peau d'orange, or skin edema of any magnitude. (Tethering or dimpling of the skin or nipple inversion should not be interpreted as skin infiltration. Patients with these conditions are eligible.)
* Ipsilateral lymph nodes that on clinical examination are found to be fixed to one another or to other structures (cN2 disease).
* Suspicious palpable nodes in the contralateral axilla or palpable supraclavicular or infraclavicular nodes, unless there is biopsy evidence that these are not involved with tumor.
* Prior therapy for breast cancer, including irradiation, chemotherapy, biotherapy, and/or hormonal therapy, with the exception of tamoxifen. Tamoxifen may be given as adjuvant therapy before study entry, but only if it was started within 28 days before randomization. Patients who started tamoxifen within 28 days before randomization and who are being considered for chemotherapy must have their tamoxifen stopped at the start of chemotherapy.
* Prior history of breast cancer, except LCIS.
* Any sex hormonal therapy, e.g., birth control pills, ovarian hormonal replacement therapy, etc. (These patients are eligible only if this therapy is discontinued prior to randomization.) Exceptions: patients may use low-dose estrogen vaginal creams or Estring® for symptomatic vaginal dryness, raloxifene (or other selective estrogen receptor modulators [SERMs]) for the prevention of osteoporosis, and luteinizing-hormone-releasing hormone (LHRH) agonists/antagonists for the purpose of medical ovarian ablation as a component of adjuvant therapy for the breast cancer.
* Patients currently taking alendronate (Fosamax®) or other bisphosphonates or calcitonin to treat or prevent osteoporosis are not eligible.
* Non-malignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude a patient from being subjected to any of the treatment options or would prevent prolonged follow-up.
* Psychiatric or addictive disorders that would preclude obtaining informed consent.
* Pregnancy or lactation at the time of proposed randomization. This protocol excludes pregnant or lactating women because the effects of clodronate on such women have not been studied fully.
* Bilateral malignancy or a mass or mammographic abnormality in the opposite breast suspicious for malignancy unless there is biopsy proof that the mass is not malignant.
* Special conditions for ineligibility of lumpectomy patients: Irradiation and surgery. The following patients will also be ineligible:

  * Patients with diffuse tumors (as demonstrated on mammography) that would not be considered surgically amenable to lumpectomy.
  * Patients treated with lumpectomy in whom there is another clinically dominant mass or mammographically suspicious abnormality within the ipsilateral breast remnant. Such a mass must be biopsied and demonstrated to be histologically benign prior to randomization or, if malignant, must be surgically removed with clear margins.
  * Patients in whom the margins of the resected specimen are involved with invasive tumor or ductal carcinoma in situ (DCIS). Additional surgical resections to obtain free margins are allowed. Patients in whom tumor is still present after the additional resection(s) must undergo mastectomy to be eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3323 (Actual)
Dates: Start 2001-01; Primary Completion 2011-03 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (17):
- United States (17):
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - Medcenter One Health System, Bismarck, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Danville Radiation Therapy Center, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - University of Washington School of Medicine, Seattle, Washington

REFERENCES:
- [Background] Ruggiero SL, Mehrotra B, Rosenberg TJ, Engroff SL. Osteonecrosis of the jaws associated with the use of bisphosphonates: a review of 63 cases. J Oral Maxillofac Surg. 2004 May;62(5):527-34. doi: 10.1016/j.joms.2004.02.004. PMID 15122554
- [Result] Atula S, Powles T, Paterson A, McCloskey E, Nevalainen J, Kanis J. Extended safety profile of oral clodronate after long-term use in primary breast cancer patients. Drug Saf. 2003;26(9):661-71. doi: 10.2165/00002018-200326090-00005. PMID 12814333
- [Result] Atula ST, Paterson AHG, Powles TJ, et al.: Safety profile of oral clodronate during long-term use in primary breast cancer patients. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-100, 25, 2003.
- [Result] Powles T, Paterson S, Kanis JA, McCloskey E, Ashley S, Tidy A, Rosenqvist K, Smith I, Ottestad L, Legault S, Pajunen M, Nevantaus A, Mannisto E, Suovuori A, Atula S, Nevalainen J, Pylkkanen L. Randomized, placebo-controlled trial of clodronate in patients with primary operable breast cancer. J Clin Oncol. 2002 Aug 1;20(15):3219-24. doi: 10.1200/JCO.2002.11.080. PMID 12149294
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- [Derived] Paterson AH, Anderson SJ, Lembersky BC, Fehrenbacher L, Falkson CI, King KM, Weir LM, Brufsky AM, Dakhil S, Lad T, Baez-Diaz L, Gralow JR, Robidoux A, Perez EA, Zheng P, Geyer CE Jr, Swain SM, Costantino JP, Mamounas EP, Wolmark N. Oral clodronate for adjuvant treatment of operable breast cancer (National Surgical Adjuvant Breast and Bowel Project protocol B-34): a multicentre, placebo-controlled, randomised trial. Lancet Oncol. 2012 Jul;13(7):734-42. doi: 10.1016/S1470-2045(12)70226-7. Epub 2012 Jun 14. PMID 22704583

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Clodronate | Arm 2: Placebo
Started | 1662 | 1661
Completed | 1655 | 1656
Not Completed | 7 | 5
Not completed — no follow up data | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Clodronate: Clodronate
- Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | Clodronate | Placebo | Total
Number analyzed (Participants) | 1662 | 1661 | 3323
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (10.5) | 53 (10.4) | 54 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1662 | 1661 | 3323
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival.
Description: Time to first event where an event is any recurrences, 2nd primary or death to determine the percentage of patients disease free at 8 years
Time Frame: 8 years
Measure: Number; unit: percentage of patients
Arm/Group | Arm 1: Clodronate | Arm 2: Placebo
Number analyzed (Participants) | 1655 | 1656
percentage of patients | 81.0 | 79.6

2. Secondary Outcome: Skeletal Metastasis Free Survival
Description: Time from randomization to first diagnosis of skeletal metastasis to determine the percentage of patient free of skeletal metastasis at 8 years
Time Frame: 8 years
Measure: Number; unit: percentage of patients
Arm/Group | Arm 1: Clodronate | Arm 2: Placebo
Number analyzed (Participants) | 1655 | 1656
percentage of patients | 95.7 | 94.6

3. Secondary Outcome: Overall Survival
Description: Time from randomization to any death to determine the percentage of patients alive at 8 years
Time Frame: 8 years
Measure: Number; unit: percentage of patients
Arm/Group | Arm 1: Clodronate | Arm 2: Placebo
Number analyzed (Participants) | 1655 | 1656
percentage of patients | 90.6 | 89.3

4. Secondary Outcome: Relapse Free Survival
Description: Time from randomization to any local, regional, or distant recurrence of breast cancer to determine the percentage of patients relapse free at 8 years
Time Frame: 8 years
Measure: Number; unit: percentage of patients
Arm/Group | Arm 1: Clodronate | Arm 2: Placebo
Number analyzed (Participants) | 1655 | 1656
percentage of patients | 89.9 | 88.3

5. Secondary Outcome: Incidence of Non-skeletal Metastasis
Description: Time from randomization to incidence of non-skeletal metastasis to determine the percentage of patients free from non-skeletal metastasis at 8 years
Time Frame: 8 years
Measure: Number; unit: percentage of patients
Arm/Group | Arm 1: Clodronate | Arm 2: Placebo
Number analyzed (Participants) | 1655 | 1656
percentage of patients | 94.8 | 93.2

ADVERSE EVENTS:
Description: Participants at Risk includes any patient who submitted an AE form.
Arm/Group | Clodronate | Placebo
All-Cause Mortality (participants affected / at risk) | 5/1612 | 12/1623
Serious Adverse Events (participants affected / at risk) | 340/1612 | 350/1623
Other Adverse Events (participants affected / at risk) | 73/1612 | 107/1623
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clodronate (N=1612) | Placebo (N=1623)
Abdominal pain (Gastrointestinal disorders) | 8 | 4
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 2 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alanine aminotransferase increased (ALT/SGPT) (Investigations) | 15 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 2
Anemia (Blood and lymphatic system disorders) | 10 | 8
Anorexia (Metabolism and nutrition disorders) | 4 | 5
Anxiety (Psychiatric disorders) | 2 | 3
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Aspartate aminotransferase increased (AST/SGOT) (Investigations) | 10 | 7
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 8
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 6 | 2
Cardiac troponin I increased (Investigations) | 1 | 0
Cardiac troponin T increased (Investigations) | 2 | 0
Cataract (Eye disorders) | 5 | 6
Catheter related infection (Infections and infestations) | 3 | 0
Cholesterol high (Investigations) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 1
Conduction disorder (Cardiac disorders) | 2 | 1
Confusion (Psychiatric disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
CPK increased (Investigations) | 2 | 0
Creatinine increased (Investigations) | 6 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 4
Depression (Psychiatric disorders) | 5 | 10
Diarrhea (Gastrointestinal disorders) | 29 | 10
Dizziness (Nervous system disorders) | 5 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 4
Dysphasia (Nervous system disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 | 13
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 2 | 0
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 5 | 0
Fatigue (General disorders) | 7 | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 4
Fever (General disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 5 | 3
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 1
Glaucoma (Eye disorders) | 2 | 0
Headache (Nervous system disorders) | 6 | 7
Hematuria (Renal and urinary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 10 | 9
Hot flashes (Vascular disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 8 | 13
Hypertension (Vascular disorders) | 11 | 14
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 7 | 3
Hyponatremia (Metabolism and nutrition disorders) | 3 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Ileus (Gastrointestinal disorders) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 27 | 28
INR increased (Investigations) | 0 | 5
Insomnia (Psychiatric disorders) | 2 | 3
Intracranial hemorrhage (Nervous system disorders) | 2 | 3
Investigations - Other, specify (Investigations) | 1 | 0
Irregular menstruation (Reproductive system and breast disorders) | 4 | 5
Ischemia cerebrovascular (Nervous system disorders) | 6 | 3
Keratitis (Eye disorders) | 1 | 0
Lipase increased (Investigations) | 4 | 0
Lymphocyte count decreased (Investigations) | 1 | 3
Memory impairment (Nervous system disorders) | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 3
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 8 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 6
Myocardial infarction (Cardiac disorders) | 6 | 4
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 7 | 6
Neuralgia (Nervous system disorders) | 4 | 1
Neutrophil count decreased (Investigations) | 73 | 107
Pain (General disorders) | 7 | 5
Palpitations (Cardiac disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 5 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 0 | 2
Peripheral ischemia (Vascular disorders) | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 7
Personality change (Psychiatric disorders) | 1 | 0
Platelet count decreased (Investigations) | 5 | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Psychosis (Psychiatric disorders) | 1 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 | 5
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 | 2
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 2 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 1
Serum amylase increased (Investigations) | 2 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 4 | 9
Syncope (Nervous system disorders) | 6 | 5
Thromboembolic event (Vascular disorders) | 18 | 30
Urinary frequency (Renal and urinary disorders) | 2 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 | 0
Vascular disorders - Other, specify (Vascular disorders) | 1 | 1
Ventricular arrhythmia (Cardiac disorders) | 2 | 1
Watering eyes (Eye disorders) | 1 | 0
Weight gain (Investigations) | 3 | 5
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Wound infection (Infections and infestations) | 17 | 17
White blood cell decreased (Investigations) | 45 | 66
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 12 | 5
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 | 5
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Visceral arterial ischemia (Vascular disorders) | 1 | 0
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
GGT increased (Investigations) | 2 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 4 | 4
Non-cardiac chest pain (General disorders) | 6 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 1 | 0
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 6 | 6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Clodronate (N=1612) | Placebo (N=1623)
Neutrophil count decreased (Investigations) | 73 | 107

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days